CLINICAL TRIAL: NCT01989494
Title: Evaluation of the Physical Activity Associated With Clinical Work in Anesthesia Residents and Attendings
Brief Title: Study of the Physical Activity in Anesthesiologists
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Vesela Kovacheva, MD, Clinical Instructor of Anesthesia, Brigham and Women's Hospital
Other Study IDs: 2013P001171
Record Dates: First submitted 2013-11-10; First posted 2013-11-21 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Healthy
Keywords: anesthesiologists; physical activity; pedometer; wellness; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Attendings: Anesthesiology Attendings who will wear a pedometer for five days while at work
  Interventions: Device: Pedometer
- CA1 Residents: Anesthesiology residents in their first year of anesthesiology residency who will wear a pedometer for five days while at work
  Interventions: Device: Pedometer
- CA2 and CA3 Residents: Anesthesiology residents in their second year of anesthesiology residency who will wear a pedometer for five days while at work

INTERVENTIONS:
Device: Pedometer — All groups will receive a pedometer to measure their daily steps
  Other Names: Pedusa PE-771 Tri-Axis Multi-Function Pocket Pedometer
  Groups: Attendings; CA1 Residents

SUMMARY:
This study will measure and compare the physical activity of the anesthesiologists during routine daily work in the operating room as determined by the pedometer-counted steps and to estimate the average daily physical activity by using a seven day exercise recall survey.

DETAILED DESCRIPTION:
This study aims to:

1. Measure and compare the physical activity of the anesthesiology residents and attendings during routine daily work in the main operating room as determined by the pedometer-counted steps walked by every individual
2. Estimate the physical activity outside of work by responding to survey of the past seven day exercise recall

The primary objective of this study is to compare the physical activity of resident and attending anesthesiologists. We hypothesize that the attendings will walk more steps than residents at work, but it is possible that the residents will be more active in their spare time. In addition, we hypothesize that the first year residents, likely associated with inefficiency in work pattern, will have more physical activity at work compared to the third year residents. The final objective of this study is to compare the physical activity of these two groups to the recommended guidelines for healthy lifestyle.

We anticipate that this study will provide us with an idea of the physical activity of the 'average anesthesiologist' in USA and will be useful for determining the need of promoting exercise for healthier lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiology residents and attendings scheduled to work in the main operating room for regular day shift who volunteer for the study

Exclusion Criteria:

* Refusal to be enrolled in the study
* Medical conditions which restrict/prohibit exercise, e.g. recent injury, recent surgical procedure, arthritis
* Pregnancy
* Part-time or on call subjects will be excluded, as well as anyone scheduled to work outside the Main Operating Room, e.g. ICU, endoscopy, obstetrics.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This is a prospective observational and retrospective survey study of the physical activity of the anesthesiologists, which would require subjects to wear pedometer in five consecutive days at work as well as recall their physical activity in the past seven-day week.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
steps walked while at work | 5 days
  We will measure the daily steps walked while at work, using a pedometer, over a period of 5 normal work days in the operating room

SECONDARY OUTCOMES:
overall level of physical activity | past 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Vesela Kovacheva, MD PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States